CLINICAL TRIAL: NCT05516706
Title: Dynamic Stretching Versus Plyometric Push up Training on Upper Body Performance in Cricketers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01021 Mahnoor
Record Dates: First submitted 2022-04-28; First posted 2022-08-25 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Sports Physical Therapy
Keywords: plyometric, dynamic stretching, agility
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: There were two groups
Who Masked: Participant
Masking Description: There were two groups one group perform dynamic stretching and the other group performed plyometric pushups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic stretching (Active Comparator): This group performed warm up and dynamic stretching exercise for six weeks.
  Interventions: Other: Plyometric push up
- Plyometric push up (Active Comparator): This group performed Warm up and plyometric push up for six weeks.
  Interventions: Other: Dynamic stretching

INTERVENTIONS:
Other: Dynamic stretching — Participants in this group performed a 10 minutes warm-up followed by 15 minutes of dynamic stretching exercises which included arm cross-over, scapular scaption, upper body twist walking lunges, cat and cow pose, and rotator cuff movements.
  Arms: Plyometric push up
Other: Plyometric push up — Participants in this group performed 10 minutes of warm-up followed by 15 minutes of plyometric push training which included one-arm push-ups and depth push up
  Arms: Dynamic stretching

SUMMARY:
A comparison of dynamic stretching and plyometric pushup training on upper body performance tests of cricketers was performed.

DETAILED DESCRIPTION:
A Randomised control trial was performed for six weeks in which a sample size of 22 was taken participants were divided into two groups in which one group performed warm-up and dynamic stretching and the other group performed warm-up plyometric pushup.

ELIGIBILITY:
Inclusion Criteria:

* Active cricket players ( who are currently laying cricket on the field)
* National-level cricket players having experience of 3 to 6 months
* Age 18 to 25 years
* Male cricketers

Exclusion Criteria:

* History of recent fracture of cervicothoracic region
* Disc prolapse stage 3
* Any other comorbid condition

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
One Arm Hop test | 6th week
  One Arm Hop test is used to measure upper body strength, power, and stability. The test is performed on both dominant and non-dominant hand. Participants begins in push up position with one hand on his back a 10.cm block was placed right next to the test arm the participant was asked to touch the block five times keeping his posture correct. The time in which they were able to complete the reps was recorded in minutes.

SECONDARY OUTCOMES:
Medicine Ball throw test | 6th week
  Medicine Ball throw test had good reliability. It is used for assessing upper body power. The participants stand with a medicine ball held in overhead position he is asked to throw as far as possible without moving his feet forward the distance in meters from standing position to the point where ball hits the ground is measured in feet.

OTHER OUTCOMES:
Y- Balance Test | 6th week
  Upper Quadrant -Y- Balance Test has a good test retest reliability. It is used to measure Upper body mobility and stability. It is performed by participants in plank position is asked to placed cones in superior lateral, inferior lateral and medial direction. The mean of distance between the cones was measured in inch's and cm for both left and right hand consecutively.

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Awan, Phd, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal Cptial, Pakistan

IPD SHARING:
Plan to Share IPD: No